CLINICAL TRIAL: NCT06477731
Title: The Effect of Waiting Time in the Premedication Room on Anxiety and Intraoperative Anesthetic Need
Brief Title: Waiting Time in the Premedication Room on Anxiety
Status: Active, not recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assoc. Prof., Istinye University
Other Study IDs: istinye erkan
Record Dates: First submitted 2024-06-22; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Total Anesthetic Consumption

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: total anesthetic consumption — total anesthetic consumption required to reach the optimal depth of anesthesia (BIS 50) depending on the anxiety of the waiting period in the preoperative waiting room and the degree of anxiety.

SUMMARY:
The primary purpose of the study is to determine the total anesthetic consumption required to reach the optimal depth of anesthesia (BIS 50) depending on the anxiety of the waiting period in the preoperative waiting room and the degree of anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age group of 18 and over
* Being literate and able to communicate
* Individuals will have surgery in ENT, Urology, Brain Surgery, Orthopedics, General Surgery, Plastic Surgery, CVS and gynecology and obstetrics departments.
* Agreeing to participate in the research voluntarily

Exclusion Criteria:

* alcohol or drug use
* history of psychiatric illness
* central nervous system disease
* use of psychotropic medication
* pregnancy
* lack of vision, hearing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 130 patients over the age of 18 who will receive general anesthesia and undergo surgical procedures will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-07-25 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
total anesthetic consumption | 1 month
  The primary purpose of the study is to determine the total anesthetic consumption required to reach the optimal depth of anesthesia (BIS 50) depending on the anxiety of the waiting period in the preoperative waiting room and the degree of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayrak A, Sagiroglu G, Copuroglu E. Effects of Preoperative Anxiety on Intraoperative Hemodynamics and Postoperative Pain. J Coll Physicians Surg Pak. 2019 Sep;29(9):868-873. doi: 10.29271/jcpsp.2019.09.868. PMID 31455484
- [Result] Ahmetovic-Djug J, Hasukic S, Djug H, Hasukic B, Jahic A. Impact of Preoperative Anxiety in Patients on Hemodynamic Changes and a Dose of Anesthetic During Induction of Anesthesia. Med Arch. 2017 Oct;71(5):330-333. doi: 10.5455/medarh.2017.71.330-333. PMID 29284900
- [Result] Maranets I, Kain ZN. Preoperative anxiety and intraoperative anesthetic requirements. Anesth Analg. 1999 Dec;89(6):1346-51. doi: 10.1097/00000539-199912000-00003. PMID 10589606